CLINICAL TRIAL: NCT00691340
Title: Systematic Characterization of the Cellular Proteome From Human Leukocytes of Glaucoma Patients in Comparison With Patients With Alzheimer's Disease
Brief Title: Cellular Proteome From Leukocytes of Glaucoma Patients in Comparison With Patients With Alzheimer's Disease
Status: Withdrawn | Type: Observational
Why Stopped: was replaced by another study. Problems with recruitment.
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University Hospital, Bonn (Other)
Responsible Party: Sponsor
Other Study IDs: 075-WUK-2008-002
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Alzheimer's Disease; Glaucoma
Keywords: POAG; Alzheimer's disease; cellular proteome; human leucocytes; vasospasm; Healthy subjects
MeSH Terms: conditions — Alzheimer Disease; Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Control 1 (young subjects)
- 2: Control 2 (old subjects)
- 3: Glaucoma patients
- 4: Alzheimer patients

SUMMARY:
Glaucoma is a worldwide leading cause of blindness. The key feature of this ocular neuropathy is characterized by an excavating optic nerve head. Loss of retinal ganglion cells is the final end point in blinding diseases of the optic nerve such as glaucoma. It is known that neuronal cell death in glaucoma occurs by an apoptotic mechanism. In earlier studies the investigators could demonstrate that the process of apoptosis is reflected in circulating leukocytes by different parameters, like differential mRNA expression and an increased fragmentation of the DNA. Such alterations point out a relationship between cellular stress and apoptotic events.

Based on the results of mRNA-expression the investigators also expect alterations on the protein level.

This study is, therefore, designed to characterize the proteome related to the proteins involved in cell death related pathways.

Thus, the expression pattern of several proteins in leukocytes from patients with primary open angle glaucoma will be analyzed by techniques like Western-blot and tandem mass spectrometry. These samples will be compared with samples from healthy controls. In addition, they will also be compared with samples from patients with Alzheimer's disease. Since glaucoma is a neurodegenerative disease, these patients will be included as positive controls in this study.

DETAILED DESCRIPTION:
Hypothesis:

Differences in the proteome concerning cell death pathways of glaucoma patients correspond to the differences in the mRNA expression of these patients.

Specific aims:

Characterization of the cellular proteome from human leukocytes of glaucoma patients compared to healthy controls and patients with Alzheimer's disease.

Background:

Glaucoma is a worldwide leading cause of blindness. The key feature of this ocular neuropathy is characterized by an excavating optic nerve head. Loss of retinal ganglion cells is the final end point in blinding diseases of the optic nerve such as glaucoma. It is known that neuronal cell death in glaucoma occurs by an apoptotic mechanism. In earlier studies we could demonstrate that this cell death is reflected in circulating leukocytes by different parameters, like differential mRNA expression, and an increased fragmentation of the DNA. The differences in mRNA expression indicate a close relationship to cellular stress conditions and apoptotic events: increased mRNA expression was detected for p53, 20S proteasome alpha subunit, ABC1 transporter, p21(WAF1/CIP1), 14-3-3 sigma factor, MMP-9 and MMP-14, and TIMP-1.

Based on the assumption that glaucoma patients may differ on the level of their expression for these mRNAs, we expect that similar differences should exist at the protein level.

This study is, therefore, designed to characterize the proteome related to the proteins involved in cell death related pathways.

ELIGIBILITY:
Inclusion Criteria:

* German native speakers
* Age between 18-85 years
* Primary open-angle glaucoma (POAG) with and without vasospasm
* An inclusion criterion for one control group is Alzheimer's disease.

Exclusion Criteria:

Any history of:

* Ocular or systemic diseases other than glaucoma or Alzheimer's disease
* Drug or alcohol abuse
* Any condition potentially interfering with the visual field results. Visual fields will be obtained from the chart.
* Mental impairment interfering with the ability to cooperate and understand the purpose of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Glaucoma patients Alzheimer's patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Selim Orguel, MD, Study Director — University Hospital, Basel, Switzerland